CLINICAL TRIAL: NCT03829358
Title: The Role of Probiotics in Improving Quality of Life in Women With Functional Constipation: Randomized Double-blind Controlled Trial
Brief Title: The Role of Probiotics in Improving Quality of Life in Women With Functional Constipation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Murdani Abdullah, Clinical Professor, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMART CITY #AID-497-A-1600004; Sub Grant #IIE-00000078-UI-1 (Other Grant/Funding Number: USAID/SHERA - SMART CITY)
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Constipation - Functional
Keywords: Constipation; Quality of Life; Probiotic; PAC-QOL
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Lactobacillus plantarum IS-10506
  Interventions: Drug: Lactobacillus plantarum IS-10506
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lactobacillus plantarum IS-10506 — Fermented milk containing probiotic Lactobacillus plantarum IS-10506 to be consumed once daily for three weeks.
  Arms: Probiotic
Drug: Placebo — Fermented milk containing placebo to be consumed once daily for three weeks.
  Arms: Placebo

SUMMARY:
This study aimed to investigate the relationship between administration of probiotics and improvement in quality of life in women with functional constipation.

ELIGIBILITY:
Inclusion Criteria:

* Being declared healthy based on initial examination and the Structured Interview Questionnaire (SIQ)
* Having the symptoms and signs of functional constipation refer to ROME IV
* Able to communicate well
* Able to consume 1 bottle of fermented milk each day for three weeks
* Not using antibiotic no later than one week before supplementation

Exclusion Criteria:

* Diagnosed with functional bowel disorder
* Using anesthesia at least 4 weeks before treatment
* Having a serious pathological disorder (carcinoma)
* During healing phase of acute gastrointestinal disorders at least 4 weeks before treatment
* Having severe heart disease
* Taking chronic medications such as antidepressants or analgesics

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2018-02-24 (Actual); Primary Completion 2018-07-21 (Actual); Study Completion 2018-07-21 (Actual)

PRIMARY OUTCOMES:
Improvement in quality of life | Three weeks after intervention.
  Improvement in quality of life were assessed using PAC-QOL© (Patient Assessment of Constipation - Quality of Life) questionnaire, consisting of four domains: physical discomfort, psychosocial discomfort, worries/concerns, and satisfaction.
  * Physical discomfort, minimum score 0, maximum score 16, lower value represents better outcome
  * Psychosocial discomfort, minimum score 0, maximum score 32, lower value represents better outcome
  * Worries/concerns, minimum score 0, maximum score 44, lower value represents better outcome
  * Satisfaction, minimum score 0, maximum score 20, higher value represents better outcome
  Total score = physical discomfort + psychosocial discomfort + worries/concerns - satisfaction
  • Total score, minimum score -20, maximum score 92, lower value represents better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Maulahela, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Puskesmas Petamburan, Jakarta, DKI Jakarta, Indonesia

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT03829358/Prot_SAP_000.pdf